CLINICAL TRIAL: NCT01176474
Title: A Phase I Trial of a Vaccine Combining Multiple Class I Peptides and Montanide ISA 51VG With Escalating Doses of Anti-PD-1 Antibody Nivolumab or Ipilimumab With Nivolumab For Patients With Resected Stages IIIC/ IV Melanoma
Brief Title: Vaccine Combining Multiple Class I Peptides and Montanide ISA 51VG With Escalating Doses of Anti-PD-1 Antibody Nivolumab or Ipilimumab With Nivolumab For Patients With Resected Stages IIIC/ IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Medarex (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15651; NCI-8316 (Other: NCI protocol #)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma | interventions — Protein Subunit Vaccines; CTAG1B protein, human; Nivolumab; spartalizumab; Antibodies; Immunotherapy; Peptides; Ipilimumab; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nivolumab and Peptide Vaccine (Experimental): Cohorts 1 through 3: Participants will receive nivolumab with the peptide vaccine within 8 days after their first apheresis procedure.
  Vaccine Combining Multiple Class I Peptides and Montanide ISA 51 VG with Escalating Doses of Anti-PD-1 Antibody Nivolumab (BMS-936558). Level 1: 1 mg/kg Nivolumab + peptide vaccine. Level 2: 3 mg/kg Nivolumab + peptide vaccine. Level 3: 10 mg/kg Nivolumab + peptide vaccine.
  Interventions: Biological: NY-ESO-1 157-165 (165V); Drug: Nivolumab; Biological: gp100:280-288 (288V); Drug: Montanide ISA 51 vegetable grade (VG); Procedure: Apheresis Procedure
- Nivolumab and Ipilimumab (Experimental): Cohorts 4 and 5. Participants will receive their first dose of nivolumab with ipilimumab within 28 days after screening blood draws. Both drugs will be given. Cohort 4: nivolumab 1mg/kg plus ipilimumab 3mg/kg. Cohort 5: nivolumab 3mg/kg plus ipilimumab 1mg/kg.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Biological: NY-ESO-1 157-165 (165V) — The vaccine contains two peptides from two different proteins (peptides are pieces that make up proteins) called gpl00 and NY-ES0-1.
  Route of Administration: When prepared as a vaccine emulsion with Montanide ISA 51 VG, the vaccine is given by deep subcutaneous injection.
  Method of Administration: The 0.5 mg vaccine emulsion dose is administered as a 1 mL injection (0.5 mg/1 mL) as a deep subcutaneous injection in the anterior thigh of the same extremity. Injections should be separated by at least 3 cm to avoid the formation of coalescent granulomas. All 4 peptides (total of 6 injections) will be administered in the same thigh and alternating thighs will be used for each subsequent treatment.
  Other Names: NSC 717388; peptide vaccine; NY-ESO-1; ESO-165V Peptide
  Arms: Nivolumab and Peptide Vaccine
Drug: Nivolumab — Nivolumab (BMS-936558) is a fully human monoclonal antibody (HuMAb) against programmed death-1 (PD-1).
  Nivolumab will be given at the following dosages: 1, 3, or 10 mg/kg.
  Nivolumab will be administered as an i.v. infusion, using a volumetric pump with a 0.2 micron in-line filter at the protocol-specified dose(s) and rate.
  Other Names: BMS-936558; NSC 748726; Anti PD-1; antibody; MDX-1106; Immunotherapy; HMA
Biological: gp100:280-288 (288V) — The vaccine contains two peptides from two different proteins (peptides are pieces that make up proteins) called gpl00 and NY-ES0-1.
  Route of Administration: When prepared as a vaccine emulsion with Montanide ISA 51 VG, the vaccine is given by deep subcutaneous injection.
  Method of Administration: The 0.5 mg vaccine emulsion dose is administered as a 1 mL injection (0.5 mg/1 mL) as a deep subcutaneous injection in the anterior thigh of the same extremity.
  Other Names: NSC 683473; Peptide; g9-288-9V Peptide
  Arms: Nivolumab and Peptide Vaccine
Drug: Montanide ISA 51 vegetable grade (VG) — Route of Administration: Administer peptide vaccine emulsions prepared with Montanide® ISA 51 VG by deep subcutaneous injection.
  Method of Administration: Divide peptide vaccine emulsion dose volumes of greater than 1.5 mL into 2 or more injections. Administer injections typically into the anterior thigh deep subcutaneous tissue. Perform subsequent injections in rotating sites. Use a 20 or 21 gauge needle for deep subcutaneous injection of the peptide vaccine emulsion.
  Other Names: NSC 737063
  Arms: Nivolumab and Peptide Vaccine
Drug: Ipilimumab — Ipilimumab will be given at the following dosage: 3 mg/kg.
  Ipilimumab will be administered as an i.v. infusion, using a volumetric pump with a 0.2 micron in-line filter at the protocol-specified dose(s) and rate.
  Other Names: NSC 732442
  Arms: Nivolumab and Ipilimumab
Procedure: Apheresis Procedure — Some blood will be removed from the participant's veins and processed by a machine to remove a small portion of the white cells. The rest of the blood will be returned into their veins. This procedure is called "apheresis." Apheresis is done to collect cells to allow the investigators to understand how their immune system is functioning before and after receiving nivolumab and vaccine. This will be done for research purposes only. The red cells and blood clotting cells will not be permanently removed during this procedure. White blood cells will need to be removed by apheresis before participants receive the study drug.
  Arms: Nivolumab and Peptide Vaccine

SUMMARY:
The purpose of this study is to test the side effects of an investigational vaccine with an immune booster, or 2 different boosters together. Investigators also want to find out its effects on the immune system and whether it will decrease the chance that melanoma will return.

DETAILED DESCRIPTION:
Up to 5 dose cohorts will be studied. Participants will be assigned to a dose cohort in the order they enter the study.

* 1 mg/kg of NIVOLUMAB + peptide vaccine (1 mg/kg cohort), then
* 3 mg/kg of NIVOLUMAB + peptide vaccine (3 mg/kg cohort), then
* 10 mg/kg of NIVOLUMAB + peptide vaccine (10 mg/kg cohort), then
* 1 mg/kg NIVOLUMAB + ipilimumab 3 mg/kg combination cohort
* 3 mg/kg NIVOLUMAB + ipilimumab 1 mg/kg combination cohort

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of resected Stages IIIC/ IV melanoma, with no evidence of disease clinically and radiologically. All melanomas regardless of primary site of disease will be allowed.
* HLA-A*0201 positive as determined by deoxyribonucleic (DNA) allele-specific polymerase chain reaction (PCR) assay; HLA restriction is not required for cohort 4
* Positive staining of most recently resected tumor tissue with antibodies to 1 or more of the following: human melanoma black 45 (HMB 45) for gp100, NY-ESO-1, and/or MART-1
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) must have been completed at least 4 weeks before study drug administration, and all adverse events have either returned to baseline or stabilized.
* Prior treated brain or meningeal metastases must be without magnetic resonance imaging (MRI) evidence of progression for at least 8 weeks and off immunosuppressive doses of systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration.
* Prior systemic radiation therapy must have been completed at least 4 weeks before study drug administration. Prior focal radiotherapy completed at least 2 weeks before study drug administration. No radiopharmaceuticals (strontium, samarium) within 8 weeks before study drug administration.
* Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before study drug administration.
* Completed nitrosourea treatment at least 6 weeks before administration of any study drug.
* Prior surgery that required general anesthesia must be completed at least 4 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration and participants should be recovered.
* Screening laboratory values must meet the following criteria: white blood cells (WBCs) ≥ 2000 cells/μL, neutrophils ≥ 1500 cells/μL, platelets ≥ 100 x 10^3/μL, hemoglobin ≥ 9.0 g/dL, serum creatinine ≤ 2 mg/dL, aspartic transaminase (AST) ≤ 2.5 x upper limit of normal (ULN) without, and ≤ 5 x ULN with hepatic metastasis, alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis, bilirubin ≤ 2 x ULN (except participants with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL).
* Females of childbearing potential (FOCBP) must: Agree to use using a reliable form of contraception (e.g., oral contraceptives, intrauterine device, double barrier method of condom and spermicidal) for at least 28 days prior to the first dose of any study drug, during the Treatment Period (and Treatment/Follow-up if receiving study drug), and for at least 70 days after the last dose of any study drug; have a negative serum β-human chorionic gonadotropin (β-HCG) at Screening.
* For female participants to be considered as not having childbearing potential, they must meet 1 or more of the following criteria: postmenopausal for at least 24 consecutive months; surgically sterile (ie, have had a hysterectomy or bilateral oophorectomy); females with irregular menstrual periods and/or on hormone replacement therapy must have a documented serum follicle stimulating hormone level > 35 mIU/mL.
* Male participants must agree to the use of male contraception during the Treatment Period and for at least 180 days after the last dose of any study drug.
* Must have read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
* Systemic hypersensitivity to Montanide ISA 51 VG or any vaccine component.
* Prior non-melanoma malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast.
* Any active autoimmune disease or documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo or resolved childhood asthma/atopy.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Positive tests for hepatitis B virus surface antigen (HBV SAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
* Prior therapy with an anti-Programmed Death-1(anti-PD-1), anti-Programmed Death-Ligand 1 (anti-PD-L1), anti-programmed death-ligand-2 (anti-PD-L2), or anti-cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody(or any other antibody targeting T cell co-stimulation pathways).
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids.
* Underlying medical condition (eg, a condition associated with diarrhea) that, in the Investigator's opinion, would make the administration of either study drug or both study drugs hazardous to the participant or obscure the interpretation of toxicity determination or adverse events.
* Pregnant or nursing.
* Current participation in another clinical study involving treatment with medications, radiation or surgery, or prior participation in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-08-13 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Time to Relapse | Start of study treatment through end of follow-up period - up to 5 years
  Scanning and exams to detect recurrence will take place periodically during treatment and follow-up until relapse is confirmed.

SECONDARY OUTCOMES:
Overall Survival (OS) | Start of study treatment until withdrawal of consent for follow-up or death - up to 6 years
  OS: Time from start of study treatment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Khushalani NI, Vassallo M, Goldberg JD, Eroglu Z, Kim Y, Cao B, Ferguson R, Monson KR, Kirchhoff T, Amato CM, Burke P, Strange A, Monk E, Gibney GT, Kudchadkar R, Markowitz J, Brohl AS, Pavlick A, Richards A, Woods DM, Weber J. Phase II clinical and immune correlate study of adjuvant nivolumab plus ipilimumab for high-risk resected melanoma. J Immunother Cancer. 2022 Nov;10(11):e005684. doi: 10.1136/jitc-2022-005684. PMID 36450385